CLINICAL TRIAL: NCT00730392
Title: "ENBREL® (Etanercept) Administration to Patients Newly Diagnosed With Type 1 Diabetes Mellitus: Feasibility-Safety Study" ("Study")
Brief Title: Etanercept in New Onset Type 1 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Teresa Quattrin, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20020197
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes, Etanercept, honeymoon period
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 drug, 2 placebo (Experimental): 1. Etanercept
  2. Placebo
  Interventions: Drug: Etanercept; Drug: Placebo

INTERVENTIONS:
Drug: Etanercept — The study drug was provided in lyophilized 10 mg vials to be reconstituted with 1 ml of diluent/vial and was administered at a dose of 0.4 mg/Kg up to maximum dose of 25 mg/dose SC twice weekly
Drug: Placebo — administered at 0.4 mg/Kg/dose SC up to 25 mg max twice weekly

SUMMARY:
The investigators hypothesized that the administration of Etanercept to children newly diagnosed with T1DM may be able to interdict the progression of T1DM. The aim of this study is to evaluate the feasibility and safety of Etanercept administration to pediatric patients recently diagnosed with type 1 DM.

DETAILED DESCRIPTION:
This is a double-blind randomized 24-week placebo-controlled feasibility and safety study. Subjects received study drug for a 24- week period, followed by 4 and 12-week wash out periods.

ELIGIBILITY:
Inclusion Criteria:

* Males and females subjects with T1DM aged 3-18 years
* Positive GAD 65 and/or islet cell antibody
* HbA1c at diagnosis above 6%
* Insulin regimen with 3 injection of insulin daily (as described below)
* White blood count between 3,000-10,000 and platelets > 100,000
* Normal ALT and AST, creatinine < 1.8 mg/dl
* T1DM duration equal or less than 4 weeks

Exclusion Criteria:

* Infection requiring IV antibiotics at diagnosis or within past 14 days from study entry
* BMI over 85th percentile for age and gender
* Unstable household
* Unable to provide compliance with study drug, insulin and study visits,
* Evidence of psychiatric disease in the potential study subject and/or primary care taker
* And chronic diseases, including additional autoimmune disorders with the exception of euthyroid autoimmune thyroiditis

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2002-10; Primary Completion 2007-10 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
The primary end points of this study are percent change from baseline for HbA1c and C-peptide area under the curve (AUC). | At baseline and at the end of the 24-week blind treatment

SECONDARY OUTCOMES:
Secondary end points are insulin dose and number of insulin injection discontinued, if any | At baseline and at end of the 24-week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Quattrin, MD, Principal Investigator — School of Medicine and Biochemical Sciences-SUNYAB

REFERENCES:
- [Derived] Mastrandrea L, Yu J, Behrens T, Buchlis J, Albini C, Fourtner S, Quattrin T. Etanercept treatment in children with new-onset type 1 diabetes: pilot randomized, placebo-controlled, double-blind study. Diabetes Care. 2009 Jul;32(7):1244-9. doi: 10.2337/dc09-0054. Epub 2009 Apr 14. PMID 19366957